CLINICAL TRIAL: NCT04528680
Title: Phase 1 / 2 Trial of Blood-brain Barrier Opening With an Implantable Ultrasound Device SonoCloud-9 and Treatment With Albumin-bound Paclitaxel and Carboplatin in Patients With Recurrent Glioblastoma
Brief Title: Ultrasound-based Blood-brain Barrier Opening and Albumin-bound Paclitaxel and Carboplatin for Recurrent Glioblastoma
Acronym: SC9/ABX
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: CarThera (Industry); Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adam M Sonabend, Assistant Professor, Feinberg School of Medicine, Neurological Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 20C03
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma; Gliosarcoma; GBM; Glioblastoma Multiforme; Glioblastoma, IDH-wildtype; Recurrent Glioblastoma
Keywords: ultrasound; SonoCloud; blood-brain barrier; paclitaxel; albumin-bound paclitaxel; Abraxane®; carboplatin
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Sonication; Drug Therapy; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- SC9/ABX (phase 1); SC9/ABX/Carboplatin (phase 2) (Experimental): Infusion of albumin-bound paclitaxel immediately followed by sonication using the SC9 device and microbubbles in order to open the blood-brain barrier in phase 1. In phase 2, patients will receive carboplatin immediately prior to sonication using the SC9 device and microbubbles in order to open the blood-brain barrier, then will receive albumin-bound paclitaxel upon completion of sonication.
  Interventions: Device: Sonication for opening of blood-brain barrier; Drug: Chemotherapy, albumin-bound paclitaxel; Drug: Chemotherapy, carboplatin

INTERVENTIONS:
Device: Sonication for opening of blood-brain barrier — Implantation of SC-9 device and repeat activation of 9 ultrasound emitters during i.v. injection of microbubbles
  Other Names: SonoCloud-9 device, SC-9
Drug: Chemotherapy, albumin-bound paclitaxel — Intravenous infusion of ABX over 30 minutes
  Other Names: Abraxane®; ABX
Drug: Chemotherapy, carboplatin — Intravenous infusion of carboplatin over 30 minutes
  Other Names: Paraplatin

SUMMARY:
Paclitaxel is among the most active agents against glioblastoma in preclinical models. However, its clinical use has been hampered by the blood-brain barrier (BBB). In this trial we will implant a novel device with 9 ultrasound emitters allowing to temporarily and reversibly open the BBB immediately prior to chemotherapy infusion with albumin-bound paclitaxel.

In the phase 1 component, increasing doses of chemotherapy will be delivered as long deemed safe based on the prior patient not experiencing severe toxicity. Once the the recommended dosing has been established, carboplatin will be added to the regimen and additional patients will be treated in order to better evaluate the antitumor efficacy of this novel treatment.

The device will be implanted at the time of surgical resection of the recurrent tumor. During that procedure and when feasible, a first test dose of the chemotherapy will be administered in the operating room after sonication (procedure of activating ultrasound and opening the BBB) and tissue concentrations in different parts of the resected tumor will be measured. In select patients, the sonication procedure may occur immediately after the test dose of chemotherapy is administered.

The objectives of this trial are to establish a safe and effective dose of albumin-bound paclitaxel, to demonstrate that the opening of the BBB increases chemotherapy concentration in the tumor, and to estimate how effective this treatment is in reducing the tumor burden and prolonging life.

DETAILED DESCRIPTION:
Eligible patients will undergo craniotomy for tumor resection. During the tumor resection and when possible, an initial low dose of albumin-bound paclitaxel will be given following sonication. In select patients, the sonication procedure may occur immediately after the test dose of chemotherapy is administered. The sonication device will be implanted at the end of the procedure. In phase 1, about two weeks after surgery, patients will undergo sonication and albumin-bound paclitaxel administration with MRI to quantify extent of blood brain barrier opening. Sonication and administration of albumin-bound paclitaxel will continue every 3 weeks until disease progression. The planned albumin-bound paclitaxel starting dose is 40 mg/m2, to be escalated in the absence of significant toxicity up to 260 mg/m2. Blood samples for circulating tumor DNA will also be collected before and after each sonication. In phase 2, pre-sonication carboplatin at AUC 5 will be added to the regimen, with a safety run-in for the first 6 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Isocitrate Dehydrogenase 1 (IDH1) wild-type glioblastoma on pathology from initial surgery (e.g. IDH R132H neg); morphologic or molecular determination of grade 4
2. Ability to undergo contrast-enhanced MRI
3. Radiographic evidence of tumor recurrence/progression after failure of 1 - 2 lines of prior therapy
4. Measurable or evaluable disease

   1. Measurable: contrast-enhancement (bidirectional diameters ≥ 1cm) on MRI
   2. Non-measurable/evaluable: contrast-enhancement diameters < 1 cm
5. Maximal tumor diameter pre-surgery ≤ 70 mm on T1wMRI
6. Candidate for at least partial surgical resection
7. Greater 12 weeks from completion of radiation therapy
8. Age ≥ 18 years
9. If receiving dexamethasone for mass effect, a stable daily dose of dexamethasone at < 6 mg within 7 days of registration, or if dexamethasone dose is decreasing, average daily dose of < 6 mg in the 7 days prior to registration. Patients on dexamethasone for reasons other than mass effect may still be enrolled.
10. WHO performance status ≤ 2 (equivalent to Karnofsky Performance Status (KPS) of ≥70)
11. Adequate hepatic, renal and bone marrow function, documented with normal laboratory values or no more than grade 1 outside the norm performed within 14 days prior to registration
12. For patients with a childbearing potential

    1. Negative pregnancy test within 14 days prior to registration
    2. Agreement to use adequate contraception for the duration of study participation, and for 3 and 6 months after the last dose of albumin-bound paclitaxel for men and women of childbearing potential, respectively.
13. Have the ability to understand and the willingness to sign a written informed consent prior to registration on study
14. Be willing and able to comply with the protocol for the duration of the study
15. Provide written, signed and dated informed consent prior to study registration. NOTE: no study-specific screening procedures may be performed until written consent has been obtained

Exclusion Criteria:

1. Have multifocal disease that cannot be encompassed in the ultrasound fields:

   1. e.g. > 70-mm apart
   2. tumor located in the posterior fossa
2. Patients at risk of cranial wound dehiscence
3. Have uncontrolled epilepsy or require treatment with enzyme-inducing antiepileptics
4. Have clinical evidence of peripheral neuropathy on examination
5. Have received any other investigational agents within 4 weeks of registration
6. Have received prior therapy with or have history of allergic reactions attributed to compounds of similar chemical or biologic composition to paclitaxel or carboplatin
7. Medical contraindications to Abraxane® or carboplatin
8. Have an uncontrolled intercurrent illness
9. Are pregnant or nursing
10. Have a history of active malignancy within 3 years prior to registration.
11. Have a known history of hypersensitivity reactions to perflutren lipid microsphere components or to any of the inactive ingredients in Definity® (the FDA-approved ultrasound contrast agent to be used in this study)
12. Patients with coils, clips, shunts, intravascular stents, and/or non-removable wafer, non resorbable dura substitute, or reservoirs.
13. Patients with medical need to continue antiplatelet therapy.
14. Patients with known significant cardiac disease, known to have right-to-left shunts, severe pulmonary hypertension (pulmonary artery pressure > 90 mmHg), uncontrolled systemic hypertension, or adult respiratory distress syndrome (patient at risk for microbubble reaction).
15. Patients with impaired thermo-regulation or temperature sensation (due to device)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (Phase1) | 1st treatment cycle = 3 weeks
  Occurrence of ≥ grade 3 treatment related toxicity
1-year survival rate (Phase 2) | 12-months
  Survival time from date of tumor resection and device implantation
Relationship between overall survival and SSR3 (Phase 2) | through study completion, an average of 2 years
  Survival time from date of tumor resection and device implantation

SECONDARY OUTCOMES:
Incidence of side effects/toxicity associated with Sonication/ABX treatment | 12 months
  Safety and tolerance

OTHER OUTCOMES:
Extent of tumor and peritumoral tissue covered by BBB opening | 1st cycle (cycle = 3 weeks)
  increase in Gd contrast enhancement post sonication
Objective response rate (RANO) | 6 months
  measurement of tumor shrinkage (if there is residual disease)
Measurement of circulating tumor DNA, methods and units for this measure are to be determined and still under evaluation. | 1st cycle, cycles 2 - 6 as applicable (cycle = 3 weeks)
  compare before and after sonication

CONTACTS AND LOCATIONS:
Overall Officials: Roger Stupp, MD, Study Chair — Northwestern University; Adam M Sonabend, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Idbaih A, Canney M, Belin L, Desseaux C, Vignot A, Bouchoux G, Asquier N, Law-Ye B, Leclercq D, Bissery A, De Rycke Y, Trosch C, Capelle L, Sanson M, Hoang-Xuan K, Dehais C, Houillier C, Laigle-Donadey F, Mathon B, Andre A, Lafon C, Chapelon JY, Delattre JY, Carpentier A. Safety and Feasibility of Repeated and Transient Blood-Brain Barrier Disruption by Pulsed Ultrasound in Patients with Recurrent Glioblastoma. Clin Cancer Res. 2019 Jul 1;25(13):3793-3801. doi: 10.1158/1078-0432.CCR-18-3643. Epub 2019 Mar 19. PMID 30890548
- [Background] Sonabend AM, Stupp R. Overcoming the Blood-Brain Barrier with an Implantable Ultrasound Device. Clin Cancer Res. 2019 Jul 1;25(13):3750-3752. doi: 10.1158/1078-0432.CCR-19-0932. Epub 2019 May 10. PMID 31076548
- [Background] Zhang DY, Dmello C, Chen L, Arrieta VA, Gonzalez-Buendia E, Kane JR, Magnusson LP, Baran A, James CD, Horbinski C, Carpentier A, Desseaux C, Canney M, Muzzio M, Stupp R, Sonabend AM. Ultrasound-mediated Delivery of Paclitaxel for Glioma: A Comparative Study of Distribution, Toxicity, and Efficacy of Albumin-bound Versus Cremophor Formulations. Clin Cancer Res. 2020 Jan 15;26(2):477-486. doi: 10.1158/1078-0432.CCR-19-2182. Epub 2019 Dec 12. PMID 31831565
- [Derived] Gould A, Luan Y, Hou Y, Korobova FV, Chen L, Arrieta VA, Amidei C, Ward R, Gomez C, Castro B, Habashy K, Zhang D, Youngblood M, Dmello C, Bebawy J, Bouchoux G, Stupp R, Canney M, Yue F, Iruela-Arispe ML, Sonabend AM. Endothelial response to blood-brain barrier disruption in the human brain. JCI Insight. 2024 Dec 26;10(4):e187328. doi: 10.1172/jci.insight.187328. PMID 39724015
- [Derived] Sonabend AM, Gould A, Amidei C, Ward R, Schmidt KA, Zhang DY, Gomez C, Bebawy JF, Liu BP, Bouchoux G, Desseaux C, Helenowski IB, Lukas RV, Dixit K, Kumthekar P, Arrieta VA, Lesniak MS, Carpentier A, Zhang H, Muzzio M, Canney M, Stupp R. Repeated blood-brain barrier opening with an implantable ultrasound device for delivery of albumin-bound paclitaxel in patients with recurrent glioblastoma: a phase 1 trial. Lancet Oncol. 2023 May;24(5):509-522. doi: 10.1016/S1470-2045(23)00112-2. PMID 37142373
- [Derived] Dmello C, Sonabend A, Arrieta VA, Zhang DY, Kanojia D, Chen L, Gould A, Zhang J, Kang SJ, Winter J, Horbinski C, Amidei C, Gyorffy B, Cordero A, Chang CL, Castro B, Hsu P, Ahmed AU, Lesniak MS, Stupp R, Sonabend AM. Translocon-associated Protein Subunit SSR3 Determines and Predicts Susceptibility to Paclitaxel in Breast Cancer and Glioblastoma. Clin Cancer Res. 2022 Jul 15;28(14):3156-3169. doi: 10.1158/1078-0432.CCR-21-2563. PMID 35552677